CLINICAL TRIAL: NCT04942964
Title: A Phase 1 Open-label Study to Evaluate the Effect of Mild and Moderate Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of ASP0367 Compared to Participants With Normal Hepatic Function
Brief Title: A Study to Evaluate ASP0367 in Participants With Mild/Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0367-CL-1102
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Hepatic Impairment; Healthy Volunteers
Keywords: Mild and moderate hepatic impairment; Liver function; ASP0367; Pharmacokinetics; MA-0211; Healthy Volunteers
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ASP0367: Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment will receive a single dose of ASP0367 under fasting conditions on day 1.
  Interventions: Drug: Bocidelpar
- ASP0367: Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment will receive a single dose of ASP0367 under fasting conditions on day 1.
  Interventions: Drug: Bocidelpar
- ASP0367: Normal Hepatic Function (Experimental): Participants with normal hepatic function will receive a single dose of ASP0367 under fasting conditions on day 1.
  Interventions: Drug: Bocidelpar

INTERVENTIONS:
Drug: Bocidelpar — Oral
  Other Names: MA-0211, ASP0367

SUMMARY:
The purpose of this study is to evaluate the effect of ASP0367 in participants with mild and moderate hepatic impairment compared to healthy participants with normal hepatic function. The study will also evaluate the safety and tolerability of ASP0367 in participants with mild and moderate hepatic impairment compared to healthy participants with normal hepatic function.

DETAILED DESCRIPTION:
The study will comprise of three groups based on hepatic function. Participants will be screened for up to 28 days prior to investigational product (IP) administration on Day 1. Eligible participants will be admitted to the clinical unit on Day -1 and will be residential for a single period of six days/five nights. On Day 1, participants will receive a single oral dose of ASP0367 under fasting conditions followed by a 96-hour in-house blood and urine sampling period. Participants are to remain semirecumbent for four hours postdose. Standard safety and tolerability assessments will be conducted. Participants will be discharged from the clinical unit on Day 5 on the condition that all required assessments have been performed and that there are no medical reasons for a longer stay in the clinical unit.

The study will be completed with an end-of-study visit (ESV). The ESV will take place five to nine days after the last pharmacokinetic sample is collected or at the time of early discontinuation from the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a BMI range of 18.5 to 36.0 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 28 days after IP administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 28 days after IP administration.
* Female participant must not donate ova starting at dose of IP and throughout the study period and for 28 days after IP administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the study period and for 28 days after IP administration.
* Male participant must not donate sperm during the study period and for 28 days after IP administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 28 days after IP administration.
* Participant agrees not to participate in another interventional study while participating in the present study.

Additional Criteria for Participants with Hepatic Impairment:

* Participant has mild (Child-Pugh classification Class A, score 5 or 6) or moderate (Child-Pugh classification Class B, score 7 to 9) hepatic impairment at screening

Exclusion Criteria:

* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to day -1.
* Participant has had a partial hepatectomy within 1 year prior to screening.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP0367 or any components of the formulation used.
* Participant has received a COVID-19 vaccine within the 2 weeks prior to IP administration or will have a COVID-19 vaccine dose before the ESV.
* Female participant who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Participant has had previous exposure with ASP0367.
* Participant has used moderate or strong inducers of CYP3A within the 3 months prior to day -1.
* Participant has used proton-pump inhibitors within the 2 weeks prior to IP administration.
* Participant has used Histamine-2 blockers within 24 hours prior to IP administration.
* Participant has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to IP administration.
* Participant has/had febrile illness or symptomatic, viral (excluding chronic hepatitis B virus and hepatitis C virus), bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Participant has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Participant is an employee of Astellas, the study-related CROs or the clinical unit.
* Participant has a positive result for SARS-CoV-2 test at screening.
* Participant has creatinine level outside normal limits on day -1. In such a case, the assessment may be repeated once.

Additional Criteria for Participants with Hepatic Impairment:

* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy not related to current disease state.
* Participant has cardiac troponin I (cTnI) > upper limit of normal (ULN) (or cardiac troponin T [cTnT]) > ULN if cTnI is not available). In such a case, the assessment may be repeated once.
* Participant has a mean pulse < 45 or > 100 bpm; mean systolic blood pressure > 160 mmHg; mean diastolic blood pressure > 100 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Participant has a mean QT interval using Fridericia's correction (QTcF) of > 460 msec for male participants and > 480 msec for female participants on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Participant who has had a change in dose regimen of medically required medication(s) in the 2 weeks prior to screening (permitted concomitant medications) and/or participant for whom dose changes are likely to occur during the study (minor dose changes are allowed in agreement with the sponsor) and/or participant has used nonpermitted concomitant medication(s) in the 3 weeks prior to admission to the clinical unit (nonpermitted concomitant medications include any known hepatic enzyme-altering agents, compounds, vitamins or natural herbal remedies, e.g., St. John's Wort known to restrict metabolism).
* Participant has a history of consuming > 14 units for male participants and > 7 units for female participants of alcoholic beverages per week within 3 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 1 year prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the participant tests positive for alcohol at screening or on day -1.
* Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or on day -1, unless the positive test is due to prescription drug use that is approved by the principal investigator and sponsor.
* Participant has a positive serology test for hepatitis A virus antibodies (IgM), hepatitis B surface antigen (HBsAg) or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening.
* Participant has fluctuating or rapidly deteriorating hepatic function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of hepatic impairment within the screening period (e.g., advanced ascites, infection of ascites, fever, active gastrointestinal bleeding).
* Participant has a presence of a hepatocellular carcinoma, or an acute liver disease caused by an infection or drug toxicity.
* Participant has severe portal hypertension or surgical portosystemic shunts, including transjugular intrahepatic portosystemic shunt.
* Participant has biliary liver cirrhosis, biliary obstruction or other cause of hepatic impairment not related to parenchymal disorder and/or disease of the liver.
* Participant has signs of significant hepatic encephalopathy (hepatic encephalopathy grade ≥ 2).
* Participant has severe ascites and/or pleural effusion.
* Participant has esophageal or gastric varices which have a high risk of clinically significant hemorrhage.
* Participant has thrombocyte level below 40 × 10^9/L and/or hemoglobin < 90 g/L.
* Participant has had previous liver transplantation.

Additional Criteria for Healthy Participants with Normal Hepatic Function:

* Participant has any of the liver function tests (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase and total bilirubin) ≥ 1 × ULN or international normalized ratio > 1.1 on day -1. In such a case, the assessment may be repeated once.
* Participant has cTnI > ULN (or cTnT > ULN if cTnI is not available) at screening.
* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Participant has any clinically significant abnormality following the physical examination, ECG and protocol-defined clinical laboratory tests at screening or on day -1.
* Participant has a mean pulse < 45 or > 90 bpm; mean SBP > 150 mmHg; mean DBP > 90 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Participant has a mean QTcF of > 430 msec for male participants > 450 msec for female participants on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Participant has used any prescribed or nonprescribed drugs (including vitamins and natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to IP administration, except for occasional use of acetaminophen (up to 2 g/day), topical dermatological products (including corticosteroid products), hormonal contraceptives and hormone replacement therapy.
* Participant has a history of consuming > 14 units for male participants and > 7 units for female participants of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the participant tests positive for alcohol at screening or on day -1.
* Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or on day -1.
* Participant has a positive serology test for HAV antibodies (IgM), hepatitis B surface antigen, HCV antibodies or antibodies to HIV type 1 and/or type 2 at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of ASP0367 in Plasma: Area Under The Concentration-time Curve From Time of Dosing Extrapolated to Time Infinity (AUCinf) | Up to 5 days
  AUCinf will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of ASP0367 in Plasma: Area Under Concentration-time Curve From Time of Dosing to the Last Measurable Concentration (AUClast) | Up to 5 days
  AUClast will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of ASP0367 in Plasma: Maximum Concentration (Cmax) | Up to 5 days
  Cmax will be recorded from the PK plasma samples collected.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Day 16
  Adverse Events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a participant, temporally associated with the use of investigational product (IP), whether or not considered related to the IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP. This includes events related to the comparator and events related to the (study) procedures.
Number of Participants with Laboratory Value Abnormalities and/or AEs | Up to Day 16
  Number of participants with potentially clinically significant laboratory values
Number of Participants with Vital Sign Abnormalities and/or AEs | Up to Day 16
  Number of participants with potentially clinically significant vital signs values.
Number of Participants With 12-lead Electrocardiogram (ECG) Abnormalities and/or AEs | Up to Day 16
  Number of participants with potentially clinically significant 12-Lead ECG values.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (3):
- United States (3):
  - Advanced Pharma CR, LLC, Miami, Florida
  - Orlando Clinical Research Center, Inc, Orlando, Florida
  - Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.